CLINICAL TRIAL: NCT03851913
Title: The Impact on Survival of Neo-adjuvant Transarterial Chemoinfusion (TAI) for Patients With Beyond Milan Criteria BCLC Stage A/B Hepatocellular Carcinoma Who Underwent Hepatectomy: A Random, Controlled, Stage III Clinical Trial
Brief Title: The Impact on Survival of Neo-adjuvant Transarterial Chemoinfusion (TAI) for Patients With Beyond Milan Criteria BCLC Stage A/B Hepatocellular Carcinoma Who Underwent Hepatectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-165-01
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): transarterial chemoinfusion (TAI) with mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
  Interventions: Procedure: TAI
- control group (No Intervention): no neo-adjuvant treatment before operation

INTERVENTIONS:
Procedure: TAI — transarterial chemoinfusion with mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
  Arms: treatment group

SUMMARY:
To compare the impact on survival of neo-adjuvant TAI for patients with beyond Milan criteria BCLC stage A/B HCC who underwent hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old and younger than 75 years;
* ECOG PS≤1;
* proven hepatocellular carcinoma according patological examination or EASL/AASLD diagnostic criteria;
* not previous treated for tumor;
* the tumor was diagnosed as BCLC stage A/B and beyond Milan criteria;
* no distant metastasis;
* the lab test could meet:

  * neutrophil count≥2.0×109/L;
  * hemoglobin≥100g/L;
  * platelet count≥75×109/L;
  * serum albumin≥35g/L;
  * total bilirubin<2-times upper limit of normal;
  * ALT<3-times upper limit of normal;
  * AST<3-times upper limit of normal;
  * serum creatine<1.5-times upper limit of normal;
  * PT≤upper limit of normal plus 4 seconds;
  * INR≤2.2;
* sign up consent.

Exclusion Criteria:

* cannot tolerate TAI or surgery;
* distant metastasis exits;
* known history of other malignancy;
* be allergic to related drugs;
* underwent organ transplantation before;
* be treated before (interferon included);
* known history of HIV infection;
* known history of drug or alcohol abuse;
* have GI hemorrhage or cardiac/brain vascular events within 30 days;
* pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 60 months
  overall survival

SECONDARY OUTCOMES:
RFS | From date of randomization until the date of recurrence, assessed up to 60 months
  recurrence-free survival
recurrence rate | 1 year, 2 year, 3 year, 5 year after surgery
  recurrence rate
PFS | From date of randomization until the date of progression, assessed up to 60 months
  progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong, China